CLINICAL TRIAL: NCT03753659
Title: IMMULAB - A Phase II Trial of Immunotherapy With Pembrolizumab in Combination With Local Ablation for Patients With Early Stage Hepatocellular Carcinoma (HCC)
Brief Title: IMMULAB - Immunotherapy With Pembrolizumab in Combination With Local Ablation in Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMULAB
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab; Pharmaceutical Preparations; Radiofrequency Ablation; Brachytherapy

STUDY DESIGN:
Intervention Model Description: Immunotherapy with pembrolizumab in combination with local ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab with local ablation (Experimental): * Pembrolizumab 200mg IV Q3W on day 1 of cycle 1 and 2
  * Radio Frequency Ablation (RFA) / Microwave Ablation (MWA) / brachytherapy or combination of TACE with RFA, MWA or brachytherapy will be performed on day 1 of cycle 3
  * Pembrolizumab 200mg IV administration 2 days after local ablation
  * Pembrolizumab 200mg IV Q3W for up to 12 months total treatment duration
  Interventions: Drug: Pembrolizumab; Procedure: Radio Frequency Ablation (RFA); Procedure: Microwave Ablation (MWA); Radiation: Brachytherapy; Drug: Transarterial Chemoembolisation (TACE)

INTERVENTIONS:
Drug: Pembrolizumab — IV infusion
  Other Names: Study treatment
Procedure: Radio Frequency Ablation (RFA) — Local ablation via RFA will be performed via ultrasound- or CT-guided placement of a needle electrode / probe penetrating into the lesion center
  Other Names: Study treatment
Procedure: Microwave Ablation (MWA) — Local ablation via MWA will be performed via ultrasound- or CT-guided placement of a needle electrode / probe penetrating into the lesion center
  Other Names: Study treatment
Radiation: Brachytherapy — Local ablation via brachythwerapy will be performed via ultrasound- or CT-guided placement of a needle electrode / probe penetrating into the lesion center
  Other Names: Study treatment
Drug: Transarterial Chemoembolisation (TACE) — According to Investigator's choice, TACE using drug eluting beads can be performed combined with RFA, MWA or brachytherapy
  Other Names: Study treatment

SUMMARY:
This is a multicenter, single arm, prospective, open-label phase II trial investigating the clinical activity of peri-interventional treatment with the anti-PD1 antibody pembrolizumab in HCC patients who are candidates for local ablation via either radiofrequency ablation (RFA) or microwave ablation (MWA) or brachytherapy or combination of TACE with RFA, MWA or brachytherapy.

DETAILED DESCRIPTION:
The multimodal approach of combining peri-interventional administration of an immune checkpoint inhibitor and local ablation via RFA / MWA / brachytherapy or combination of TACE with RFA, MWA or brachytherapy harbors the potential to satisfy the unmet need for an improvement in the outcomes of HCC patients treated with RFA / MWA/ brachytherapy or combination of TACE with RFA, MWA or brachytherapy. Furthermore, early clinical data indicates that the combination of immune checkpoint inhibition with RFA, MWA or brachytherapy displays an acceptable safety profile, resulting in a positive benefit-risk ratio of this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of HCC
2. Has a Child-Pugh Classification score ≤ 6 for assessed liver function within 7 days before allocation (Appendix 4: Child-Pugh Score)
3. Candidate for local ablation (via either RFA or MWA or brachytherapy or combination of TACE with RFA, MWA or brachytherapy [ablation technique according to Investigator's choice]), i.e.:

   According to Investigator's assessment an R0 state can be obtained after a maximum of two RFA/MWA interventions (initial ablation + one additional re-ablation at maximum).
4. Patients (including high risk patients) with: :

   * Presence of ≤ 5 tumor nodules with diameters ≤ 7cm [longest axis] each OR
   * Vascular infiltration
5. Has received no prior systemic therapy for HCC NOTE: Patients who have received prior local therapy by transarterial chemoembolization (TACE) are not excluded if TACE has been performed >8 weeks before study allocation.
6. Have measurable disease based on RECIST 1.1. Lesions situated in a previously treated (e.g. irradiated or subject to TACE) area are considered measurable if vital tumor has been demonstrated by contrast enhanced imaging in such lesions*.
7. Male/female participants who are at least 18 years of age on the day of signing informed consent will be enrolled in this study.
8. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.

   A male participant with female partner of childbearing potential is eligible to participate if he agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
9. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
10. Have provided archival tumor tissue sample or newly obtained biopsy of a tumor lesion not previously irradiated for mandatory pre-treatment evaluation (baseline).

    * Newly obtained biopsies are preferred to archived tissue (archived specimen ≤6 months may be acceptable).
    * Core or excisional biopsies mandatory (fine needle aspiration and bone metastasis samples are not acceptable).
    * Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
    * If submitting unstained cut slides, newly cut slides should be submitted to the central pathology lab within 14 days from the date slides are cut.
    * Availability of baseline tumor biopsy samples has to be ensured by site before first dose of study medication is administered.
    * Specimens have to be sent to central pathology lab for accompanying research project.
11. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
12. Have adequate organ function as defined in the following table. Specimens must be collected within 7 days prior to the start of study treatment.

    Adequate Organ Function Laboratory Values

    Hematological
    * Absolute neutrophil count (ANC) ≥1500/µL
    * Platelets ≥100 000/µL
    * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L(a)

    Renal

    - Creatinine OR ≤1.5 × Upper Limit of Normal (ULN) OR Measured or calculated(b) creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN

    Hepatic
    * Total bilirubin ≤2.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >2.5 × ULN
    * aspartate aminotransferase [AST (SGOT)] and alanine aminotransferase [ALT (SGPT)] ≤5 × ULN

    Coagulation

    - International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
13. If patient has concurrent Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection, meets the following criteria:

    * Patients with HBV or HCV infection should be monitored for viral levels during study participation.
    * Patients with detectable hepatitis B surface antigen (HBsAg) or detectable HBV DNA should be managed per local treatment guidelines. Controlled (treated) hepatitis B subjects will be allowed if they started treatment at the time point of enrollment into the study by the latest and treatment is continued during study participation.
    * Patients with detectable HCV RNA are usually not treated for their HCV infection. However, patients treated for HCV are considered suitable for inclusion if antiviral therapy has been completed prior to first administration of study drug.

Exclusion Criteria:

1. Extrahepatic disease
2. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
3. Presence of tumor thrombus involving main trunk of portal vein
4. Has at Screening and/or has had any prior history of Grade ≥ 2 hepatic encephalopathy
5. Has at Screening pericardial effusion, uncontrollable pleural effusion, or clinically significant ascites defined as meeting either of (a) detectable ascites on Screening physical examination OR (b) has at Screening ascites requiring paracentesis
6. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
7. Has received prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-Programmed death-ligand 1 (anti-PD-L1), or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, Cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), OX 40, CD137).
8. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or at least 5 half-lives of the respective drug/IMP (whichever is longer) prior to allocation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
9. Has received prior radiotherapy within 4 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
10. Has received a live vaccine within 4 weeks or for a period of at least 5 half-lives of the respective drug/IMP (whichever is longer) before Screening and during Screening for this trial prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
11. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks or for a period of at least 5 half-lives of the respective drug/IMP (whichever is longer) before Screening and during Screening for this trial.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks or at least 5 half-lives of the respective drug/IMP (whichever is longer) after the last dose of the previous investigational agent.
12. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
13. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
14. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
15. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
16. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
17. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
18. Has an active infection requiring systemic therapy (exception: HBV infection - see inclusion criteria).
19. Has a history of Human Immunodeficiency Virus (HIV) (mandatory testing for HIV during screening is required).
20. Has a known history of active tuberculosis(Bacillus Tuberculosis).
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
24. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 | After 6 weeks (2 cycles) of treatment
  Evaluation of ORR according to RECIST 1.1 after two cycles of pembrolizumab and before performing local ablation will allow testing of the hypothesis that pre-interventional treatment with pembrolizumab before local ablation will result in conversion / downstaging of borderline candidates for local ablation. Furthermore, ORR is generally accepted as a valid endpoint for efficacy evaluation in one-armed trials without control group.

SECONDARY OUTCOMES:
Time to recurrence (TTR) according to RECIST 1.1 | 18 months of Follow Up
  TTR and recurrence free survival, have meanwhile been accepted by medicinal agencies in drug approval processes as they allow for quicker efficacy assessment. This is most important in explorative clinical trials in early phases (like this phase II trial) as it allows for more rapid evaluation of the potential of new treatment approaches. Furthermore, many of these parameters are not influenced by follow-up therapies.
Recurrence free survival according to RECIST 1.1 | 18 months of Follow Up
  TTR and recurrence free survival, have meanwhile been accepted by medicinal agencies in drug approval processes as they allow for quicker efficacy assessment. This is most important in explorative clinical trials in early phases (like this phase II trial) as it allows for more rapid evaluation of the potential of new treatment approaches. Furthermore, many of these parameters are not influenced by follow-up therapies.
Overall survival (OS) | 18 months of Follow Up
  Overall survival will be evaluated and is still considered the gold standard for efficacy evaluation in clinical trials. Its major drawback is the potentially long observation period necessary for OS evaluation - especially in the curative setting as represented by the treatment approach in this trial.
Incidence and severity of adverse events | 12 months of treatment + 18 months of Follow Up
  Incidence and severity of adverse events according to the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Identification of molecular biomarkers in tumor tissue and blood samples by immunohistochemical and molecular analyses in a central lab | 9 weeks of treatment
  Correlation analyses between selected molecular parameters and clinical data to identify molecular biomarkers like PD-1, PD-L1 and PD-L2) and immune cell infiltrates (like e.g. IGHM, CD3, CD8, FOXP3, CD68, CD205) as well as chemokines (CXCL9. CXCL10, CXCL13) and invasion markers (MMP7, MMP9) in tumor tissue and blood samples predictive for ORR, TTR, recurrence free survival and OS. Analyses will be performed by immunohistochemical and molecular methods in a central lab.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — IKF Klinische Krebsforschung GmbH atKrankenhaus Nordwest
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.